CLINICAL TRIAL: NCT03058354
Title: Retrospective Study to Investigate Total Intravenous Anaesthesia (TIVA) With Propofol on Postoperative Pain and Side Effects After Surgery
Brief Title: Study to Investigate TIVA With Propofol on Postoperative Pain and Side Effects
Status: Withdrawn | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW17-001
Record Dates: First submitted 2017-02-07; First posted 2017-02-20 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Anesthesia, General

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group TIVA: Patient undergoing surgery at Queen Mary Hospital, Hong Kong between 2014 to 2016 using intraoperative TIVA with propofol.
  Interventions: Drug: Propofol
- Group GA: Patient undergoing surgery at Queen Mary Hospital, Hong Kong between 2014 to 2016 using general anaesthesia methods other than intraoperative TIVA with propofol.
  Interventions: Procedure: general anaesthesia

INTERVENTIONS:
Drug: Propofol — Patient undergoing surgery at Queen Mary Hospital, Hong Kong between 2014 to 2016 using intraoperative TIVA with propofol.
  Groups: Group TIVA
Procedure: general anaesthesia — Patient undergoing surgery at Queen Mary Hospital, Hong Kong between 2014 to 2016 using general anaesthesia methods other than intraoperative TIVA with propofol.
  Groups: Group GA

SUMMARY:
Propofol is a commonly used anaesthetic with rapid recovery and less side effects and total intravenous anaesthesia (TIVA) with propofol is a common technique now. The reduction on certain serum pro- inflammatory cytokines may lead to more smooth post- surgical recovery.

Recent case report proved the analgesic effect of propofol infusion. However other animal and clinical studies showed controversial result.

The aim of this retrospective study is to investigate the postoperative analgesic effects and side effects of intraoperative TIVA with propofol in patient undergoing surgery at Queen Mary Hospital, Hong Kong between 2014 to 2016.

DETAILED DESCRIPTION:
Objectives:

1. To investigate the analgesic effects of propofol.
2. To evaluate the effect of propofol on postoperative adverse events.

Methods:

Retrospective audit.

Data Collection:

1. Demographic data;
2. Types of analgesic techniques;
3. Type of pain relief modalities;
4. Pain score up to 72 hours postoperatively;
5. Postoperative opioid consumption;
6. Incidence of adverse events during APS care;
7. Patients' satisfaction on pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthetic records and acute pain service records of patient undergone surgery between 2014 to 2016 in Queen Mary Hospital would be retrieved from the computer.

Exclusion Criteria:

* Essential data were missing.
* Patient participating in other research projects.
* Changes in postoperative pain management technique.
* Patients could not be assessed post-operatively for pain (i.e. post-operative IPPV)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery at Queen Mary Hospital, Hong Kong between 2014 to 2016.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
pain score | up to postoperative day 3
  pain score using numeral rating scale

SECONDARY OUTCOMES:
analgesic consumption | up to postoperative day 3
  analgesic consumption base on patient drug record

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No